CLINICAL TRIAL: NCT01074632
Title: A Phase 1, Open-Label Study to Determine the Effect of Calories and Fat Content on the Pharmacokinetics of Repeated Dose Lurasidone 120 mg in Subjects With Schizophrenia, Schizoaffective Disorder, or Schizophreniform Disorder.
Brief Title: Effect of Calories and Fat Content on the Pharmacokinetics of Lurasidone HCl
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: D1050267
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Schizophrenia, Schizoaffective Disorder, or Schizophreniform Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Lurasidone Hydrochloride

INTERVENTIONS:
Drug: Lurasidone HCl

SUMMARY:
The objective of this study is to evaluate the effect of calorie and fat content on the pharmacokinetics of Lurasidone HCl in subjects with schizophrenia, schizoaffective disorder, or schizophreniform disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 18 to 65 years of age
* BMI >= 19.5 and <= 37 kg/m2
* No clinically relevant abnormal laboratory values

Exclusion Criteria:

* History or presence of renal or hepatic insufficiency
* Participated in a clinical trial in the past 30 days
* Use of con meds that prolong the QT/QTc taken within 14 days prior to study drug administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - California Clinical Trials, Glendale, California
  - Clinical Research Institute, Wichita, Kansas